CLINICAL TRIAL: NCT03640325
Title: The Promoting Resilience in Stress Management (PRISM) Intervention: a Multi-site Randomized Controlled Trial for Adolescents and Young Adults Receiving Hematopoietic Cell Transplantation
Brief Title: The PRISM Intervention for Adolescents and Young Adults Receiving Hematopoietic Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Children's Hospital Los Angeles (Other); St. Jude Children's Research Hospital (Other); University of Alabama at Birmingham (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Abby Rosenberg, Associate Professor, Pediatrics, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001077 (SC-N126); R01CA225629 (NIH)
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Bone Marrow Neoplasms; Anxiety; Depression; Quality of Life; Adherence, Medication; Coping Skills; Adolescent Behavior
MeSH Terms: conditions — Neoplasms; Bone Marrow Neoplasms; Anxiety Disorders; Depression; Medication Adherence; Adolescent Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRISM (Promoting Resilience in Stress Management) (Experimental): Resilience Skills Training
  Interventions: Behavioral: PRISM (Promoting Resilience in Stress Management)
- Usual Care (No Intervention): Usual psychosocial care (control arm, no intervention)
- Caregivers (No Intervention): Caregivers of participants, no intervention

INTERVENTIONS:
Behavioral: PRISM (Promoting Resilience in Stress Management) — Manualized Skills-Training Program targeting resilience resources: stress-management, goal-setting, cognitive reframing, and meaning-making
  Arms: PRISM (Promoting Resilience in Stress Management)

SUMMARY:
Multisite Randomized Controlled Trial (RCT) testing the efficacy of the Promoting Resilience in Stress Management (PRISM) intervention among Adolescents and Young Adults receiving hematopoietic cell transplantation for hematology malignancy.

DETAILED DESCRIPTION:
The experience of hematopoietic cell transplantation (HCT) for malignancy or cancer predisposition among Adolescents and Young Adults (AYAs) is particularly difficult because age-related developmental challenges of identity, relationships, and vocation may add to the burden of cancer. Compared to other age-groups, AYAs have poorer psychosocial outcomes including increased anxiety and depression and poorer adherence to oral immunosuppressive medications. These outcomes may, in turn, predispose AYAs to disease-related morbidity and mortality such as graft-versus-host disease (GVHD) and/or cancer-relapse. A potential barrier to improving these experiences may be that AYAs have few opportunities to develop the personal resources needed to handle adversity. We have previously developed the "Promoting Resilience in Stress Management" (PRISM) intervention for AYAs with serious illness. This manualized, brief intervention is delivered in 4, 30-60 minute, one-on-one sessions, followed by a Parent/ Caregiver/ Spouse/ significant other inclusive meeting. It targets skills in stress-management and mindfulness, goal-setting, positive reframing, and meaning-making. All of these skills are associated with improved patient well-being in other populations, and preliminary findings from a recently closed phase II randomized controlled trial among AYAs with newly diagnosed cancer suggest PRISM is associated with improved health-related quality of life. This study will build on our prior experience and fill a critical knowledge gap regarding PRISM's impact among AYAs receiving HCT. Thus, we will conduct a multi-site randomized controlled trial with the primary trial outcome of patient-reported symptoms of anxiety and depression. Secondary and exploratory outcomes will include the cost-effectiveness of the intervention in this population, the impact of the intervention on parent well-being, and patient adherence to oral graft-versus-host-disease medications. We hypothesize that AYAs who receive PRISM will report fewer mixed affective symptoms, while their parents report improved quality of life and psychological distress. We also anticipate the intervention will positively impact adherence and be cost-effective. In sum, this study offers an opportunity to expand the body of knowledge regarding methodologically rigorous and evidence-based psychosocial interventions and standards of care for AYAs with hematologic malignancies. Ultimately, this research has the potential to reduce the burden of cancer in these vulnerable populations.

ELIGIBILITY:
Inclusion Criteria for adolescent/young adult (AYA) patient:

* Patient aged 12-24 years
* Receiving hematopoietic cell transplantation (HCT) for malignancy or cancer predisposition syndrome
* Within 4 weeks of HCT "day zero"
* Able to speak English
* Able to read English or Spanish
* Cognitively able to participate in interviews

Exclusion Criteria for AYA patient:

* Patient refusal
* Cognitively or physically unable to participate in interviews
* Unable to speak English
* Unable to read English or Spanish

For enrolled caregivers of AYA patient (no age limit):

Inclusion criteria:

* AYA Child of caregiver agreed to participate
* One caregiver per patient-caregiver dyad
* Parent/guardian cognitively and physically able to participate
* Parent/guardian is able to speak/read English or Spanish

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby R Rosenberg, MD, MS, MA, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital Cancer and Blood Disorders Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
All IPD will be protected and maintained by the study team

REFERENCES:
- [Derived] Taylor MR, Cole SW, Bradford MC, Zhou C, Fladeboe KM, Knight JM, Baker KS, Yi-Frazier JP, Rosenberg AR. Resilience Intervention Improves Stress-Related Gene Expression in Adolescent and Young Adult HCT Recipients. Transplant Cell Ther. 2024 Dec;30(12):1209.e1-1209.e7. doi: 10.1016/j.jtct.2024.09.014. Epub 2024 Sep 19. PMID 39303988
- [Derived] Fladeboe KM, Scott S, Comiskey L, Zhou C, Yi-Frazier JP, Rosenberg AR. The Promoting Resilience in Stress Management (PRISM) intervention for adolescents and young adults receiving hematopoietic cell transplantation: a randomized controlled trial protocol. BMC Palliat Care. 2022 May 19;21(1):82. doi: 10.1186/s12904-022-00966-9. PMID 35585525

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregiver: Caregiver of adolescent/young adult participant - surveys only no intervention.
Period: Overall Study
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care | Caregiver
Started | 50 | 44 | 49
Completed | 37 | 33 | 28
Not Completed | 13 | 11 | 21
Not completed — Withdrawal by Subject | 4 | 1 | 0
Not completed — Lost to Follow-up | 4 | 5 | 21
Not completed — Death | 5 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Caregiver data should not be considered in the comparisons or TOTAL column - those only represent the PRISM and Usual Care groups. They did not complete the same baseline measures as the PRISM and Usual Care groups so those fields are left blank for the relevant groups.
Groups:
- Caregiver: Caregiver of the adolescent/young adult participant (no intervention)
- Total: Total of all reporting groups
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care | Caregiver | Total
Number analyzed (Participants) | 50 | 44 | 49 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (4.2) | 17.1 (4.2) | 45.5 (7.5) | 16.7 (4.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 30 | 23 | 33 | 86
  Male | 20 | 21 | 7 | 48
  Missing | 0 | 0 | 9 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 33 | 23 | 30 | 86
  Hispanic | 10 | 12 | 0 | 22
  Non-Hispanic Black | 4 | 5 | 2 | 11
  Asian | 1 | 4 | 2 | 7
  Other | 2 | 0 | 2 | 4
  Missing | 0 | 0 | 13 | 13
Hospital Anxiety and Depression Scale - Total Score [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) - total score assesses anxiety and depression combined. The total score is reported here: this score is the sum of the 14 total items in this scale, 7 of which assess anxiety and 7 assess depression. Each item is scored from 0-3 which results in a total score range of 0-42. Higher scores indicate higher anxiety/depressive symptoms. Population: Caregivers were not assessed.
  units on a scale
    number analyzed (Participants) | 50 | 44 | 0 | 94
    (all) | 10.6 (5.9) | 11.4 (7.2) |  | 11.0 (6.5)
Hospital Anxiety and Depression Scale - Depression Subscale [Mean (Standard Deviation); unit: units on a scale] — 7 questions for depression, each scored on a Likert scale 0-3 for a total range of 0-21 per subscale. Higher scores indicate higher depression. Population: Caregiver group not assessed.
  units on a scale
    number analyzed (Participants) | 50 | 44 | 0 | 94
    (all) | 4.7 (3.2) | 5.2 (3.8) |  | 4.9 (3.5)
Hospital Anxiety and Depression Scale-Anxiety Subscale [Mean (Standard Deviation); unit: units on a scale] — 7 questions for anxiety, each scored on a Likert scale 0-3 for a total range of 0-21 per subscale. Higher scores indicate higher anxiety. Population: Caregiver group not assessed.
  units on a scale
    number analyzed (Participants) | 50 | 44 | 0 | 94
    (all) | 6.0 (3.3) | 6.2 (3.8) |  | 6.1 (3.8)
Snyder Hope Scale [Mean (Standard Deviation); unit: units on a scale] — Scored with a range of 0-64, higher scores imply greater levels of hopeful thought patterns. Population: Caregiver group not assessed.
  units on a scale
    number analyzed (Participants) | 50 | 44 | 0 | 94
    (all) | 47.7 (9.2) | 47.1 (9.4) |  | 47.4 (9.3)
Connor-Davidson Resilience Scale [Mean (Standard Deviation); unit: units on a scale] — 10-item measure ranging from 0-40, with higher scores indicated higher perceived resilience. Population: Caregiver group not assessed.
  units on a scale
    number analyzed (Participants) | 50 | 44 | 0 | 94
    (all) | 27.3 (6.8) | 27.5 (7.3) |  | 27.4 (7.0)
Pediatric Quality of Life - Cancer Module [Mean (Standard Deviation); unit: units on a scale] — Scored on a 0-100 scale with higher scores representing better health-related quality of life. Population: Caregiver group not assessed.
  units on a scale
    number analyzed (Participants) | 50 | 44 | 0 | 94
    (all) | 69.8 (12.6) | 68.2 (17.3) |  | 69.1 (15.9)
Generalized Anxiety Disorder Screener (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — This is a 7-item survey used to identify generalized anxiety disorder. Each item is scored on a Likert scale, with higher scores representing more anxiety. Score range is 0-21. Population: Only caregiver group assessed on this measure.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 49 | 49
    (all) |  |  | 8.1 (5.9) | 8.1 (5.9)
Patient Health Questionnaire - 8 [Mean (Standard Deviation); unit: units on a scale] — Only caregiver group assessed on this measure. This is a 8-item measure used to assess depressive symptoms. The range is 0-27 with higher scores indicated higher depression severity. Population: Only caregiver group assessed on this measure.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 49 | 49
    (all) |  |  | 6.3 (5.1) | 6.3 (5.1)
Medical Outcomes Study Rand 36-item Health Survey [Mean (Standard Deviation); unit: units on a scale] — This survey assesses generic health-related quality of life for adults. This score ranges from 0-100 with higher scores indicating better health status. Population: Only caregiver group assessed on this measure.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 49 | 49
    (all) |  |  | 71.0 (16.9) | 71.0 (16.9)

OUTCOME MEASURES:

1. Primary Outcome: Hospital Anxiety & Depression Scale (HADS) Score - Depression Sub-score
Description: The Hospital Anxiety and Depression Scale -Depression sub scale assesses mixed affective symptoms in patients with serious illness. The scale consists of 7 questions for depression. Each is scored from 0-3, for a total range of 0-21 points. "Caseness" of depression is defined as ≥8 points, with sensitivity/specificity of 0.8/0.8 for depression. The depression sub-scale will be measured as a continuous variable. Higher scores indicate more symptoms.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care
Number analyzed (Participants) | 37 | 33
score on a scale | 4.55 (3.35) | 4.03 (3.83)

2. Secondary Outcome: PedsQL Generic Core and Cancer-Related Quality of Life Score
Description: The PedsQL 4.0 Generic and 3.0 Cancer Module include 50 items evaluating health-related quality of life of adolescents and young adults (AYAs) with cancer. Items are rated on a 5-point Likert scale and total scores transformed to a 0-100 scale with higher scores representing better HRQOL. Internal consistency ranges from 0.75 to 0.92.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care
Number analyzed (Participants) | 37 | 33
score on a scale | 73.48 (14.46) | 77.14 (16.48)

3. Secondary Outcome: Connor-Davidson Resilience Scale
Description: The Connor-Davidson Resilience Scale (CD-RISC) measures inherent resiliency. The 10-item instrument has high internal consistency. Each item consists of a 5-point Likert scale (scored from zero to four). ranging from 0-40 with higher scores reflecting greater perceived resilience.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care
Number analyzed (Participants) | 37 | 33
score on a scale | 27.65 (6.95) | 29.64 (8.94)

4. Secondary Outcome: Hope Scale Scores
Description: The Snyder "Hope" Scale measures "the overall perception that one's goals can be met." The instrument scored on an 8-point Likert scale (score range 0-64). Higher scores imply greater levels of hopeful thought patterns.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care
Number analyzed (Participants) | 37 | 33
score on a scale | 47.21 (11.78) | 49.37 (10.15)

5. Secondary Outcome: Hospital Anxiety & Depression Scale Score - Anxiety Sub-score
Description: The Hospital Anxiety and Depression Scale - Anxiety sub scale assesses mixed affective symptoms in patients with serious illness. It consists of 7 questions on a 3 point Likert scale for a total range of 0-21. Higher scores indicate higher anxiety.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care
Number analyzed (Participants) | 37 | 33
score on a scale | 5.86 (3.39) | 5.13 (4.19)

6. Secondary Outcome: Generalized Anxiety Disorder Screener (GAD7)
Description: 7-item survey used to assess anxiety symptoms. Scored from 0-21 with higher scores indicated higher anxiety.
Time Frame: 6-months
Population: Only caregivers assessed for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care | Caregiver
Number analyzed (Participants) | 0 | 0 | 28
units on a scale |  |  | 5.3 (4.9)

7. Secondary Outcome: Patient Health Questionnaire-8
Description: 8-item survey assessing depression severity. Each item scored on a 4-point Likert scale with a range of 0-27. Higher scores indicate higher depression.
Time Frame: 6-months
Population: Only caregivers assessed for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care | Caregiver
Number analyzed (Participants) | 0 | 0 | 28
units on a scale |  |  | 4.5 (4.7)

8. Secondary Outcome: Medical Outcomes Study Rand 36-item Health Survey
Description: This is a measure of health-related quality of life. Scores range from 0-100 and higher scores indicate better health status
Time Frame: 6-months
Population: Only caregivers assessed for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care | Caregiver
Number analyzed (Participants) | 0 | 0 | 28
units on a scale |  |  | 72.0 (16.2)

ADVERSE EVENTS:
Time Frame: 6-months
Description: Note: no adverse events were collected for caregiver arm.
Arm/Group | PRISM (Promoting Resilience in Stress Management) | Usual Care
All-Cause Mortality (participants affected / at risk) | 5/50 | 5/44
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/44
Other Adverse Events (participants affected / at risk) | 0/50 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT03640325/Prot_SAP_000.pdf